CLINICAL TRIAL: NCT03314090
Title: Clinical Evaluation of Silicone Gel in the Treatment of Cleft Lip Scars
Brief Title: Silicone Gel in the Treatment of Cleft Lip Scars
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102-4719b
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Cleft Lip
Keywords: Cleft lip; Scar; Silicone sheet; Silicone gel
MeSH Terms: conditions — Cleft Lip; Cicatrix | interventions — Silicone Gels

STUDY DESIGN:
Intervention Model Description: Testing silicone gel in the treatment of upper lip scar
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Silicone Gel Group (Experimental): Intervention: Silicone gel (Dermatix Ultra, Menarini, Singapore) was applied twice per day (BID). The amount being similar in size to a grain of rice.
  Interventions: Drug: Silicone Gels

INTERVENTIONS:
Drug: Silicone Gels — silicone gel (Dermatix Ultra, Menarini, Singapore) was applied twice per day. The amount used being similar in size to a grain of rice.
  Other Names: Dermatix Ultra

SUMMARY:
Cleft lip / palate is the most common craniofacial anomaly in humans. Lip repair is one of the most important reconstructions for these patients, and is performed at around 3 months of age. Although the cheiloplasty scar is unavoidable and permanent, every possible measure should be considered to optimize its functional and aesthetic outcome, since the scar can be a lifelong social stigma of a cleft lip operation. Hypertrophic scarring can highlight the scar even further, and is a recognized negative outcome for cheiloplasty. Moreover, with an incidence as high as 36.3% , hypertrophic scars are more common in Asian-Orientals compared to Caucasians.

The population treated at investigator's institution is almost entirely Oriental (Taiwanese). Patients' intrinsic higher risk of hypertrophic scarring has led investigators continuously to try to improve scar quality for them. In 2011, investigator started a double-blinded, randomized, vehicle-controlled, prospective clinical trial to evaluate whether the injection of botulinum toxin A into the orbicularis oris muscle could improve the quality of the cleft lip scar . The results revealed that botulinum toxin injections into the subjacent orbicularis oris muscle produced narrower cheiloplasty scars, but provided no additional benefits in terms of scar pigmentation, vascularity, pliability or height. During that study, the parents of 14% (4/29) of the babies within the control group reported that participant baby had tried, albeit unsuccessfully, to ingest the silicone sheet at night. This caused investigator to question the safety of silicone sheeting on the upper lip in babies.

Silicone is known to be effective for treating and/or preventing hypertrophic scarring . Silicone gel has been shown to prevent hypertrophic scars in median sternotomy wounds 8. Investigators therefore conducted this clinical trial to evaluate whether post-operative use of silicone gel was non-inferior to silicone sheet for preventing hypertrophy of unilateral cleft lip repair scars.

DETAILED DESCRIPTION:
The control group consisted of 29 patients who were recruited and became controls for a previous study (Botulinum Toxin to Improve Results in Cleft Lip Repair; IRB No 101-3009C) who were treated using the current established protocol for scar care following cheiloplasty 2. This involved microporous tape placed across both cheeks and spanning the upper lip during daytime, and silicone sheets fixed with a shorter length of microporous tape (that did not span the cheeks) at night. This continued strictly for 6 months.

The Study group consisted of another 33 consecutive age-matched patients with unilateral cleft lip, whose postoperative scar care was exactly the same except the silicone sheet was replaced with silicone gel (Dermatix Ultra, Menarini, Singapore), which was applied twice per day. The parents (or caregivers) were instructed to apply silicone gel (the amount being similar in size to a grain of rice) along the upper lip scar from the nostril base to the vermillion, avoiding the wet mucosa.

Inclusion criteria were: 1. Baby born with cleft lip planned for primary lip repair around 3 months of age, . Written informed consent for the study provided by the parent/guardian. Exclusion criteria were: 1. presence of other craniofacial anomalies; 2. lack of signed informed consent from the parent/guardian.

ELIGIBILITY:
Inclusion Criteria:

* Baby born with cleft lip planned for primary lip repair around 3 months of age,
* Written informed consent for the study provided by the parent/guardian

Exclusion Criteria:

* presence of other craniofacial anomalies;
* lack of signed informed consent from the parent/guardian.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
Vacouver scar scale | Six months after surgery
  Pigmentation: 0 normal; 1 hypopigmentation; 2 Hyperpigmentation Vascularity: 0 normal; 1. pink; 2. red; 3. purple Pliability: 0 normal; 1. supple, flexible with minimal resistance; 2. Yielding, giving way to pressure; 3. firm, inflexible, not easily moved, resistant to manual pressure; 4. banding, rope-like tissue that blanches with extension of the scar; 5. contracture, permanent shortening of the scar producing deformity or distortion.
  Height: 0. normal; 1. less than 2 mm; 2. less than 5 mm; 3. more than 5 mm The sum of each item give the total scores. The score range from 0-13; with minimum of 0 being the best scar and maximum13 the worst scar
Visual Analogue Scale | Six months after surgery
  VAS with 10 grades: 0 represented the worst possible scar outcome and 10 the best possible scar outcome.
Scar width | Six months after surgery
  A standard frontally oriented photograph was taken with a surgical ruler placed on the lower lip at the six-month follow up clinic. The scar width measurements were obtained from the photographs (using the surgical ruler as the reference) by two independent raters and means calculated. A commercial photograph program for scar width measurement was utilized (Photoshop CS5 extended version 12.0; Adobe Systems Inc, San Jose, California). Scars were measured at two points: the First Point was 1 mm above the white roll; the Second Point was 1 mm below the C-flap suture line.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Chun Shin, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lin TM, Lin TY, Chou CK, Lai CS, Lin SD. Application of microautologous fat transplantation in the correction of sunken upper eyelid. Plast Reconstr Surg Glob Open. 2014 Dec 5;2(11):e259. doi: 10.1097/GOX.0000000000000141. eCollection 2014 Nov. PMID 25506542
- [Background] Chang CS, Wallace CG, Hsiao YC, Chang CJ, Chen PK. Botulinum toxin to improve results in cleft lip repair: a double-blinded, randomized, vehicle-controlled clinical trial. PLoS One. 2014 Dec 26;9(12):e115690. doi: 10.1371/journal.pone.0115690. eCollection 2014. PMID 25541942
- [Background] Chang CS, Wallace CG, Hsiao YC, Chang CJ, Chen PK. Botulinum toxin to improve results in cleft lip repair. Plast Reconstr Surg. 2014 Sep;134(3):511-516. doi: 10.1097/PRS.0000000000000416. PMID 25158709
- [Background] Chernoff WG, Cramer H, Su-Huang S. The efficacy of topical silicone gel elastomers in the treatment of hypertrophic scars, keloid scars, and post-laser exfoliation erythema. Aesthetic Plast Surg. 2007 Sep-Oct;31(5):495-500. doi: 10.1007/s00266-006-0218-1. PMID 17700980
- [Background] Signorini M, Clementoni MT. Clinical evaluation of a new self-drying silicone gel in the treatment of scars: a preliminary report. Aesthetic Plast Surg. 2007 Mar-Apr;31(2):183-7. doi: 10.1007/s00266-005-0122-0. PMID 17171514
- [Background] Kim S, Choi TH, Liu W, Ogawa R, Suh JS, Mustoe TA. Update on scar management: guidelines for treating Asian patients. Plast Reconstr Surg. 2013 Dec;132(6):1580-1589. doi: 10.1097/PRS.0b013e3182a8070c. PMID 24281584
- [Background] Borgognoni L. Biological effects of silicone gel sheeting. Wound Repair Regen. 2002 Mar-Apr;10(2):118-21. doi: 10.1046/j.1524-475x.2002.00205.x. No abstract available. PMID 12028528